CLINICAL TRIAL: NCT03693352
Title: Effect of Positive End-expiratory Pressure on Functional Residual Capacity Measured by Volumetric Capnography in Mechanically Ventilated Patients
Brief Title: Functional Residual Capacity Measured by Capnography in Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Hospital Privado de Comunidad de Mar del Plata (Other)
Responsible Party: Sponsor
Other Study IDs: 2919/1728/18
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing surgeries: Patients ASA 1-3, undergoing different types of general anesthesia that need postural changes like Trendelenburg and anti-Trendelenburg positioning.

SUMMARY:
Changes in body position during anesthesia can alter functional residual capacity and gas exchange. The monitoring of such changes in functional residual capacity is difficult at the bedside. The present study was designed to determine if volumetric capnography can detect changes in the functional residual capacity during surgery.

DETAILED DESCRIPTION:
This is a prospective and observational study designed to test the reliability of the capnodynamic equation to determine changes in functional residual capacity measured during anesthesia. The investigators will studied 40 mechanically ventilated patients undergoing general anesthesia. Functional residual capacity will be continuously measured in a non invasive way using expired carbon dioxide. Changes in functional residual capacity with standard modification in body positioning (Trendelenburg or anti-Trendelenburg position) and ventilatory settings wiil be tested.

ELIGIBILITY:
Inclusion Criteria:

* Written Inform Consent
* Programmed surgery
* Laparoscopic surgery
* Supine position

Exclusion Criteria:

* Emergency surgery
* Chronic respiratory disease
* Active smoking

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing general anesthesia for laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Functional Residual Capacity Measured by Capnography in Ventilated Patients | 6 hours
  Measurement of functional residual capacity with capnography with body positioning changes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Tusman, MD, Principal Investigator — Hospital Privado de Comunidad de Mar del Plata
Locations (1):
- Hospital Privado de Comunidad, Mar del Plata, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albu G, Wallin M, Hallback M, Emtell P, Wolf A, Lonnqvist PA, Gothberg S, Petak F, Habre W. Comparison of static end-expiratory and effective lung volumes for gas exchange in healthy and surfactant-depleted lungs. Anesthesiology. 2013 Jul;119(1):101-10. doi: 10.1097/ALN.0b013e3182923c40. PMID 23571638
- [Derived] Tusman G, Wallin M, Acosta C, Santanera B, Portela F, Viotti F, Fuentes N, Hallback M, Suarez-Sipmann F. Positive end-expiratory pressure individualization guided by continuous end-expiratory lung volume monitoring during laparoscopic surgery. J Clin Monit Comput. 2022 Oct;36(5):1557-1567. doi: 10.1007/s10877-021-00800-2. Epub 2021 Dec 29. PMID 34966951